CLINICAL TRIAL: NCT02446886
Title: Adrenocorticotropic Hormone (ACTH) Effects on Myelination in Subjects With MS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1405015090
Record Dates: First submitted 2015-05-07; First posted 2015-05-18 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; RRMS; SPMS; ACTH
MeSH Terms: conditions — Multiple Sclerosis | interventions — Adrenocorticotropic Hormone; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- One Time Treatment (Active Comparator): MS patients enrolled in this study will be randomized into:
  Intervention for Group A: 80 units/day ACTH (H.P. Acthar®)for 3-5 days (The dose could be adjusted based on the individual needs of the patients up to 80-120 units daily for 2-3 weeks.)
  Interventions: Drug: Adrenocorticotropic hormone (ACTH) gel (H.P. Acthar®)
- Monthly Treatments (Experimental): Intervention for Group B: 80 units/day ACTH (H.P. Acthar®) for 3-5 days (The dose could be adjusted based on the individual needs of the patients up to 80-120 units daily for 2-3 weeks.), followed by monthly 80 units/day ACTH for 3 days for 12 months of treatment.
  Interventions: Drug: Adrenocorticotropic hormone (ACTH) gel (H.P. Acthar®)

INTERVENTIONS:
Drug: Adrenocorticotropic hormone (ACTH) gel (H.P. Acthar®) — Adrenocorticotropic hormone (ACTH) gel, a long-acting formulation of the full sequence ACTH that includes other pro-opiomelanocortin (POMC) peptides, is considered an alternative to corticosteroids in the treatment of relapses (currently FDA approved for this indication).
  ACTH (H.P. Acthar®) gel exerts direct anti-inflammatory and immune-modulating effects within the CNS, specifically on infiltrating macrophages and resident microglia as well as protecting mature oligodendrocytes from inflammation-related damage and excitotoxicity. These effects are mediated not only via induction of endogenous corticosteroid production but also via effects on melanocortin receptors.
  Other Names: ACTH; H.P. Acthar®

SUMMARY:
The primary objective of this study is to determine if monthly pulse doses of a three-day course ACTH (H.P. Acthar®) is more effective at recovering myelin at 12 months, as measured by myelin water fraction (MWF), in new multiple sclerosis lesions as compared to one course of treatment.

The main secondary objective is to utilize every three month MWF measurements to determine the peak time of remyelination in new multiple sclerosis lesions when followed over the course of 12 months.

DETAILED DESCRIPTION:
This pilot study proposal is designed to perform a chronological measurement of MWF in new contrast-enhancing lesions in subjects treated with ACTH during an acute exacerbation of MS.

The initial course of ACTH (H.P. Acthar®) will be administered as recommended in the package insert, a subcutaneous daily dose of 80-120mg units daily for 2-3 weeks. However, as recommended in the package insert, the dosage may be individualized according to the medical condition of each subject. Therefore, the frequency and dose of the drug may be determined by considering the severity of the disease and the initial response of the subject. The typical dosing for an MS exacerbation is 80mg/day for 3-5 days and it is expected that this will be the initial dosing for the majority of thesubjects.

MS subjects enrolled in this study will be randomized into:

One Time Treatment: 80mg/day ACTH for 3-5 days (The dose could be adjusted based on the individual needs of the subjects up to 80-120mg units daily for 2-3 weeks.)

Monthly Treatments: 80mg/day ACTH for 3-5 days (The dose could be adjusted based on the individual needs of the the subjects up to 80-120mg units daily for 2-3 weeks.), followed by monthly 80 mg/day ACTH for 3 days for up to 12 months of treatment.

The Judith Jaffe Multiple Sclerosis Center currently has over 1000 subjects in a clinical and MRI database. The subjects who have signed consent for the database will have their standard of care MRI scans monitored for new enhancing lesions; this will only have to be repeated if initial scan is not completed at our MS center with our current clinical protocol. All RRMS subjects with new enhancing lesions will be considered for the study and approached regarding participation subjects that are considered candidates and consent for the study, subjects will then be randomized (1:1) to receive one course of ACTH followed by monthly pulses vs. receiving only one course of ACTH treatment. All subjects will have follow-up MRI¿s are 3 months, 6 months and 12 months post lesion onset for a total of 3 additional scans. If a patient is identified as having an enhancing lesion from MRI scan not obtained through our database, an additional scan will be obtained through the study and serve as the baseline MRI. All subjects will receive the first course of ACTH within 4 weeks of new lesion detection.

Multiple sclerosis (MS) is a very dynamic disease both biologically and clinically, which is characterized by a temporally complex pattern of inflammation, demyelination/remyelination, and axonal loss. The cycle of demyelination and remyelination has been shown to occur in MS lesions (1,2). High dose corticosteroids have been a mainstay of treatment for MS relapses. Corticosteroid treatment shortens time to recovery from relapses, presumably at least in part due to their anti-inflammatory effects. Despite their anti-inflammatory properties, corticosteroids have been shown to impair and delay remyelination in animal models of MS (3,4) and there is little clinical evidence of a longer-term beneficial effect. Adrenocorticotropic hormone (ACTH) gel, a long-acting formulation of the full sequence ACTH that includes other pro-opiomelanocortin (POMC) peptides, is considered an alternative to corticosteroids in the treatment of relapses (currently FDA approved for this indication). ACTH gel exerts direct anti-inflammatory and immune-modulating effects within the central nervous system (CNS). These effects are mediated not only via induction of endogenous corticosteroid production but also via effects on melanocortin receptors (5). Studies have shown that ACTH and other melanocortins may reduce neuroinflammatory responses (6), and ACTH has been shown to protect mature oligodendrocytes from inflammation-related damage and excitotoxicity (7). Currently however, there is a paucity of studies using more advanced MRI metrics to determine if ACTH may have reparative and neuroprotective properties in subjects with MS. We propose to study monthly courses of ACTH in subjects with new lesions and compared to the one-time treatment course of ACTH for new activity. We hypothesize that continued exposure to the anti-inflammatory effects of ACTH on new lesions would be superior to promoting remyelination as compared to a one-time treatment course. Given that the majority of endogenous remyelination is felt to begin within months after lesion development and likely to be most prominent in the few months following, a one year study is most likely sufficient to measure this process.

T2 relaxometry is a MR imaging technique in which a series of T2-weighted images at different echo times are obtained and the contribution of water associated with myelin and other tissue compartments can be differentiated using T2 decay curve analysis(8). The relative contribution of the myelin water, represented as the myelin water fraction (MWF), has been shown to highly correlate with histological myelin measurement in animal models (9) and ex-vivo brain (10,11), and has been applied to MS the subjects (12). The histological correlation of T2 relaxometry with myelin content makes it an excellent candidate as a biomarker for myelin content and it has been found to be reproducible and sensitive marker to change over time (13-16). Through the application a multi-slice 2D T2prep spiral gradient echo (GRE) imaging, T2 data can be efficiently acquired (17,18) and we have further optimized a 3D T2prep GRE sequence at 3T for which full brain coverage can be achieved within 10 minutes (19). One of the main advantages of using T2 relaxometry and MWF as a surrogate for myelin over other advanced MR modalities lies in the T2 spectrum (the T2 decay curve analysis). Both MWF and the extracellular T2 component (the intermediate peak) within the T2 spectrum) can increase with edema (20), thus once the extracellular pool stabilizes, we can ensure that any change in MWF is a true reflection of myelination.

The primary objective of this study is to determine if monthly pulse doses of a three-day course ACTH (H.P. Acthar®) is more effective at recovering myelin at 12 months, as measured by MWF, in new multiple sclerosis lesions as compared to one course of treatment.

The main secondary objective is to utilize every three-month MWF measurements to determine the peak time of remyelination in new multiple sclerosis lesions when followed over the course of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RRMS or SPMS with new contrast-enhancing lesions who will start as part of their standard of care ACTH.

Exclusion Criteria:

* Patients having received oral or IV corticosteroids within one month prior to initial scan demonstrating contrast enhancing lesion
* Patients with known or new allergy to ACTH
* Patients being treated with Natalizumab, Rituximab, and Cyclophosphamide
* Patients unwilling to have serial MRI exams
* Patients unable to undergo MRI imaging because of having an artificial heart valve, metal plate, pin, or other metallic objects in their body or is unable to complete all the MRI scans required for this study
* Patients with acute or chronic renal disease in whom administration of gadolinium may pose risk of nephrogenic systemic fibrosis
* Patients that are pregnant
* Premenopausal woman not willing to use at least one form of contraception
* Patients with a known history of diabetes mellitus
* Patients with a known history of osteoporosis or bone density values in the osteoporosis range at screening
* Progressive neurological disorder other than RRMS or SPMS
* Clinically significant cardiovascular disease, including myocardial infarct within last 6 months, unstable ischemic heart disease, congestive heart failure, or angina
* Subjects on chronic steroid therapy for treatment of MS or other systematic disease
* Subject currently has a significant medical condition (other than MS) including the following: neurological, psychiatric, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular (including uncontrolled hypertension), gastrointestinal, urological disorder, or central nervous system (CNS) infection that would pose a risk to the subject if they were to participate in the study or that might confound the results of the study

  o Note: Active medical conditions that are minor or well-controlled are not exclusionary if, in the judgment of the Primary Investigator, they do not affect risk or the subject or the study results.
* Subject is unable to cooperate with any study procedures, unlikely to adhere to the study procedures and keep appointments, in the opinion of the Investigator, or was planning to relocate during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Gauthier, DO, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- One Time Treatment: MS patients enrolled in this study will be randomized into:
  Intervention for Group A: 80 units/day ACTH (H.P. Acthar®)for 3-5 days (The dose could be adjusted based on the individual needs of the patients up to 80-120 units daily for 2-3 weeks.)
  Adrenocorticotropic hormone (ACTH) gel (H.P. Acthar®): Adrenocorticotropic hormone (ACTH) gel, a long-acting formulation of the full sequence ACTH that includes other pro-opiomelanocortin (POMC) peptides, is considered an alternative to corticosteroids in the treatment of relapses (currently FDA approved for this indication).
  ACTH (H.P. Acthar®) gel exerts direct anti-inflammatory and immune-modulating effects within the CNS, specifically on infiltrating macrophages and resident microglia as well as protecting mature oligodendrocytes from inflammation-related damage and excitotoxicity. These effects are mediated not only via induction of endogenous corticosteroid production but also via effects on melanocortin receptors.
- Monthly Treatments: Intervention for Group B: 80 units/day ACTH (H.P. Acthar®) for 3-5 days (The dose could be adjusted based on the individual needs of the patients up to 80-120 units daily for 2-3 weeks.), followed by monthly 80 units/day ACTH for 3 days for 12 months of treatment.
  Adrenocorticotropic hormone (ACTH) gel (H.P. Acthar®): Adrenocorticotropic hormone (ACTH) gel, a long-acting formulation of the full sequence ACTH that includes other pro-opiomelanocortin (POMC) peptides, is considered an alternative to corticosteroids in the treatment of relapses (currently FDA approved for this indication).
  ACTH (H.P. Acthar®) gel exerts direct anti-inflammatory and immune-modulating effects within the CNS, specifically on infiltrating macrophages and resident microglia as well as protecting mature oligodendrocytes from inflammation-related damage and excitotoxicity. These effects are mediated not only via induction of endogenous corticosteroid production but also via effects on melanocortin recep
Period: Overall Study
Arm/Group | One Time Treatment | Monthly Treatments
Started | 8 | 7
Completed | 6 | 3
Not Completed | 2 | 4
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Monthly Treatments: Intervention for Group B: 80 units/day ACTH (H.P. Acthar®) for 3-5 days (The dose could be adjusted based on the individual needs of the patients up to 80-120 units daily for 2-3 weeks.), followed by monthly 80 units/day ACTH for 3 days for 12 months of treatment.
  Adrenocorticotropic hormone (ACTH) gel (H.P. Acthar®): Adrenocorticotropic hormone (ACTH) gel, a long-acting formulation of the full sequence ACTH that includes other pro-opiomelanocortin (POMC) peptides, is considered an alternative to corticosteroids in the treatment of relapses (currently FDA approved for this indication).
  ACTH (H.P. Acthar®) gel exerts direct anti-inflammatory and immune-modulating effects within the CNS, specifically on infiltrating macrophages and resident microglia as well as protecting mature oligodendrocytes from inflammation-related damage and excitotoxicity. These effects are mediated not only via induction of endogenous corticosteroid production but also via effects on melanocortin receptors.
- Total: Total of all reporting groups
Arm/Group | One Time Treatment | Monthly Treatments | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (8.9) | 40.6 (13.4) | 37.75 (11.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Myelin Water Fraction (MWF) Within New Enhancing Lesions Over the Course of 12 Months
Description: Primary outcome: The absolute change in lesion MWF (over our test-retest variability) between baseline and one year MRI's will be calculated and compared between treatment groups.
  Method to assess lesion MWF: FAST-T2 is a multi-compartment T2 relaxometry MRI technique wherein the contribution of water associated with myelin and other tissue compartments is differentiated using T2 decay curve analysis. The relative contribution of the myelin water with respect to total water is represented as MWF. A higher MWF within a lesion reflects higher myelin content within that lesion.
  For this analysis, MWF maps were reconstructed from FAST-T2 MRI data by using a multi-voxel nonlinear least-squares data-fitting algorithm with spatial smoothness constraints. MWF was calculated as the ratio of the myelin water signal to the total water signal within a voxel. Lesion MWF is an average of the voxels present within an individual lesion.
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: myelin water fraction
Arm/Group | One Time Treatment | Monthly Treatments
Number analyzed (Participants) | 8 | 7
myelin water fraction | 1.7 (1.8) | -0.20 (1.3)
Statistical Analysis 1: Comparison: One Time Treatment vs Monthly Treatments; Previously published reproducibility of our MWF imaging (FAST-T2) has been established to be +/- 2.0 Our hypothesis for this study was the monthly ACTH would lead to greater remylination in acute MS lesions. However, to reach this goal, improvement must be beyond established reproducibility. Note: Since MWF is a fraction of myelin water to total water, it does not have a unit; Test type: Superiority; p = 0.04, t-test, 2 sided; Mean Difference (Final Values) = 1.65

2. Secondary Outcome: Physical Disability as Measured by EDSS
Description: Expanded Disability Status Scale (EDSS)
  0 Normal neurological exam, no disability in any FS 1.0 No disability, minimal signs in one FS 1.5 No disability, minimal signs in more than one FS 2.0 Minimal disability in one FS 2.5 Mild disability in one FS or minimal disability in two FS 3.0 Moderate disability in one FS, or mild disability in three or four FS. No impairment to walking 3.5 Moderate disability in one FS and more than minimal disability in several others. No impairment to walking 4.0 Significant disability but self-sufficient and up and about some 12 hours a day. Able to walk without aid or rest for 500m 4.5 Significant disability but up and about much of the day, able to work a full day, may otherwise have some limitation of full activity or require minimal assistance. Able to walk without aid or rest for 300m
  10.0 Death due to MS
  A higher score means a worse outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | One Time Treatment | Monthly Treatments
Number analyzed (Participants) | 8 | 7
score on a scale | .5 (.9) | 1.1 (1.5)

3. Secondary Outcome: Change in T2 Lesion Volume
Description: The change in T2 lesion volume between baseline and one year MRI's will be calculated and compared between treatment groups.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millimeters cubed
Arm/Group | One Time Treatment | Monthly Treatments
Number analyzed (Participants) | 8 | 7
millimeters cubed | 683.59 (1241.92) | 1092.08 (1513.45)

4. Secondary Outcome: Cortical Volume
Description: Change in cortical volume of the brain over 12 months.
Time Frame: 12 Months
Population: Data was not collected due to patient withdrawal. Too small of a sample size.
Arm/Group | One Time Treatment | Monthly Treatments
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Whole Brain Volume
Description: Change in whole brain volume over 12 months.
Time Frame: 12 months
Population: Data was not collected due to patient withdrawal. Too small of a sample size.
Arm/Group | One Time Treatment | Monthly Treatments
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Longitudinal Assessment of MWF
Description: Outcome measure: Longitudinal assessment of MWF (every 3 months) to determine the dynamics of myelin change over 12 months.
  Method to assess lesion MWF: FAST-T2 is a multi-compartment T2 relaxometry MRI technique wherein the contribution of water associated with myelin and other tissue compartments is differentiated using T2 decay curve analysis. The relative contribution of the myelin water with respect to total water is represented as MWF. A higher MWF within a lesion reflects higher myelin content within that lesion.
  For this analysis, MWF maps were reconstructed from FAST-T2 MRI data by using a multi-voxel nonlinear least-squares data-fitting algorithm with spatial smoothness constraints. MWF was calculated as the ratio of the myelin water signal to the total water signal within a voxel. Lesion MWF is an average of the voxels present within an individual lesion.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: myelin water fraction
Arm/Group | One Time Treatment | Monthly Treatments
Number analyzed (Participants) | 8 | 7
myelin water fraction | 1.7 (1.8) | -.2 (1.3)
Statistical Analysis 1: Comparison: One Time Treatment vs Monthly Treatments; Linear mixed-effects models were implemented to assess the variables of interest (lesion MWF) among patients randomized to once versus the monthly ACTH treatment group. The modeling strategy accounts for multiple lesions per patient, repeated measurements (longitudinal analysis) and the following covariates were always considered: patient age, gender, disease duration, individual T2w lesion volume, time on disease modifying treatments (DMT) prior to enrollment, and DMT during the study; Test type: Superiority; p = 0.077, Mixed Models Analysis; Mean Difference (Final Values) = 1.65; Linear mixed-effects models were implemented

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | One Time Treatment | Monthly Treatments
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2015-10-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT02446886/Prot_000.pdf